CLINICAL TRIAL: NCT02833233
Title: A Pilot Study of Pre-Operative, Single-Dose Ipilimumab, Nivolumab and Cryoablation in Early Stage/Resectable Breast Cancer
Brief Title: A Study of Pre-Operative Treatment With Cryoablation and Immune Therapy in Early Stage Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-495
Record Dates: First submitted 2016-07-12; First posted 2016-07-14 (Estimated); Results first posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer
Keywords: Early stage; Resectable; Ipilimumab; Nivolumab; Cryoablation; 16-495
MeSH Terms: conditions — Breast Neoplasms | interventions — Cryosurgery; Ipilimumab; Nivolumab

ARMS (1):
- Cryoablation and Immune Therapy (Experimental): Patients will undergo breast biopsy with cryoablation 7-10 days prior to the planned surgery, and ipilimumab with nivolumab administration 1-5 days before cryoablation. All patients will undergo surgery at the pre-determined day defined at the initial surgical consultation. Women will receive ipilimumab and nivolumab 1-5 days prior to US or MRI-guided core biopsy and cryoablation date. Intravenous ipilimumab will be administered as a single 1 mg/kg dose to be infused intravenously over 90 minutes. Intravenous nivolumab will be administered as a single 3 mg/kg dose to be infused intravenously over 60 minutes.
  Interventions: Procedure: Cryoablation; Drug: Ipilimumab; Drug: Nivolumab

INTERVENTIONS:
Procedure: Cryoablation
Drug: Ipilimumab
Drug: Nivolumab

SUMMARY:
This study is being done to evaluate the safety of combining two strategies called "cryoablation" and "immune therapy" in women with curable early stage breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Women age 18 years or older
* Confirmed histologic diagnosis of invasive adenocarcinoma of the breast, including MSKCC pathology confirmation
* ER, PR and HER2 testing in progress (i.e. on outside or MSKCC biopsy report)

  * HER2-positive pathology is permitted
* Operable tumor measuring ≥1.5 cm in maximal diameter

  * Any nodal status
  * Multifocal and multicentric disease is permitted
  * Synchronous bilateral invasive breast cancer is permitted
  * The tumor should be more than 5 mm from the skin
* No indication of distant metastases
* Breast surgery planned
* Tumor amenable to cryoablation as determined by radiologist
* ECOG performance status score of 0 or 1
* Screening laboratory values must meet the following criteria:

  * White blood cells (WBCs) ≥ 2000/μL
  * Absolute neutrophil count (ANC) ≥ 1500/μL
  * Platelets ≥ 100 x 10^3/μL
  * Hemoglobin ≥ 11.0 g/dL
  * Serum creatinine ≤ 2 mg/dL (or glomerular filtration rate ≥ 40 ml/min)
  * AST ≤ 2.5 x upper limit of normal (ULN)
  * ALT ≤ 2.5 x ULN
  * Bilirubin within normal limits (except subjects with Gilbert's syndrome, who must have total bilirubin < 3.0 mg/dL)
  * Negative HIV screening test
  * Negative screening tests for Hepatitis B and Hepatitis C. Patients with positive results that do not indicate true active or chronic infection may enroll after discussion and consensus agreement by the treating physician and principal investigator.
* Women of childbearing potential (WOCBP) must be using an acceptable method of contraception to avoid pregnancy throughout the study and for at least 3 months after the last dose of ipilimumab in such a manner that the risk of pregnancy is minimized. See below for the definition of WOCBP.
* WOCBP must have a negative serum pregnancy test within 14 days prior to the first dose of ipilimumab/nivolumab
* Women must not be breastfeeding
* Willing to adhere to the study visit schedule and the prohibitions and restrictions specified in this protocol.

Exclusion Criteria:

* Inflammatory breast cancer
* Medical history and concurrent diseases

  * Subjects with active, known or suspected autoimmune disease. Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
  * Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the subject to receive protocol therapy, or interfere with the interpretation of study results.
* Prohibited Treatments and/or Therapies

  * Chronic use of immunosuppressants and/or systemic corticosteroids (used in the management of cancer or non-cancer-related illnesses). However, use of corticosteroids is allowed for the treatment of immune related Adverse Events (irAEs), or adrenal insufficiency.
  * Any non-oncology vaccine therapy used for prevention of infectious diseases within 4 weeks prior to first dose of ipilimumab.
  * Prior treatment with a CD137 agonist, ipilimumab or other CTLA4 inhibitor;
  * Prior investigational agents within 2 weeks prior to first dose of ipilimumab;
  * Prior therapy with any anti-cancer agents including chemotherapy, adjuvant chemotherapy, immunosuppressive agents, surgery or radiotherapy within 2 weeks prior to first dose of ipilimumab.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2024-06-07 (Actual); Study Completion 2024-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Comen, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cryoablation and Immune Therapy
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cryoablation and Immune Therapy
Number analyzed (Participants) | 5
Age, Continuous [Median (Full Range); unit: years] | 54 [50 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Evaluated for Adverse Events
Description: Safety will be evaluated for all treated subjects using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events v4.0 (CTCAE).
Time Frame: 12 weeks after ipilimumab/nivolumab administration.
Measure: Count of Participants; unit: Participants
Arm/Group | Cryoablation and Immune Therapy
Number analyzed (Participants) | 5
Participants | 5

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Cryoablation and Immune Therapy
All-Cause Mortality (participants affected / at risk) | 1/5
Serious Adverse Events (participants affected / at risk) | 1/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cryoablation and Immune Therapy (N=5)
Death NOS (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cryoablation and Immune Therapy (N=5)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4
Alanine aminotransferase increased (Investigations) | 3
Hyperthyroidism (Endocrine disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 3
Alkaline phosphatase increased (Investigations) | 2
Fatigue (General disorders) | 2
Aspartate aminotransferase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Breast pain (Reproductive system and breast disorders) | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dry eye (Eye disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Hot flashes (Vascular disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Insomnia (Psychiatric disorders) | 1
Pain (General disorders) | 1
Palpitations (Cardiac disorders) | 1
Paresthesia (Nervous system disorders) | 1
Platelet count decreased (Investigations) | 1
Urinary urgency (Renal and urinary disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
White blood cell decreased (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-03): https://cdn.clinicaltrials.gov/large-docs/33/NCT02833233/Prot_SAP_000.pdf